CLINICAL TRIAL: NCT03530670
Title: The Effect of Three Different Interventions on Preoperative Anxiety in Children
Brief Title: Effect of Premedication Type on Preoperative Anxiety in Children
Acronym: EPPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bahar SAKIZCI UYAR, MD, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 42/05
Record Dates: First submitted 2018-04-18; First posted 2018-05-21 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Preoperative Anxiety
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Crossover assignment Effect of pharmacological and nonpharmacological premedication on anxiety
Who Masked: Participant
Masking Description: single (participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral midazolam (demizolam) (Active Comparator): To prevent preoperative anxiety patient premedicated by 0.5 mg/kg oral midazolam.
  In the preoperative holding area, in the operating room, while anesthesia induction by m-YPAS ( modified the Yale Preoperative Anxiety Scale) To make easier anesthesia induction While anesthesia induction by Mask Acceptance Scale
  Interventions: Other: oral midazolam
- http://www.animaturk.com/animasyon/suko-ameliyat-oluyor. (Active Comparator): To prevent preoperative anxiety by watching a short movie ( at http://www.animaturk.com/animasyon/suko-ameliyat-oluyor.) In the preoperative holding area, in the operating room, while anesthesia induction by m-YPAS ( modified the Yale Preoperative Anxiety Scale) To make easier anesthesia induction While anesthesia induction by Mask Acceptance Scale
  Interventions: Other: Film http://www.animaturk.com/animasyon/suko-ameliyat-oluyor.
- playing smartphone game (Active Comparator): To prevent preoperative anxiety by playing smartphone game ( angry birds, subway surfers, snail Bob) In the preoperative holding area, in the operating room, while anesthesia induction by m-YPAS ( modified the Yale Preoperative Anxiety Scale) To make easier anesthesia induction While anesthesia induction by Mask Acceptance Scale
  Interventions: Other: Playing smartphone game

INTERVENTIONS:
Other: oral midazolam — 0.5 mg/kg oral midazolam administered 20 minutes before anesthesia induction
  Other Names: demizolam
  Arms: oral midazolam (demizolam)
Other: Film http://www.animaturk.com/animasyon/suko-ameliyat-oluyor. — Patients will be watched a short movie (at URL:
  http://www.animaturk.com/animasyon/suko-ameliyat-oluyor.html#.Wd-YhFu0PIU) 20 minutes before induction.
  Arms: http://www.animaturk.com/animasyon/suko-ameliyat-oluyor.
Other: Playing smartphone game — Patients will be played with smartphone (angry birds, subway surfers or snail Bob) 20 minutes before induction
  Arms: playing smartphone game

SUMMARY:
Compare the effects of pharmacological and nonpharmacological premedications on preoperative anxiety and mask acceptance after adenotonsillectomy

DETAILED DESCRIPTION:
Compare the effects of 0.5 mg/kg oral midazolam, watching film 'Suko is being operated' animation film http://www.animaturk.com/animasyon/suko-ameliyat-oluyor.html#.Wd-YhFu0PIU , playing smartphone game ( subway surfers, snail Bob or angry birds) on preoperative anxiety by m-YPAS in the holding area, in the operating room and while induction of anesthesia.

Investigators also evaluated mask acceptance by Mask Acceptance Scale Investigators also evaluated post operative delirium by PAED (postanesthetic emergency delirium) scale at PACU at arrive and every 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Elective surgery

Exclusion Criteria:

* Chronic diseases
* Development disability
* Prematurity
* Neurological diseases
* Psychoactive medication use
* Hearing/visual impairment
* History of surgery

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in preoperative anxiety | Before premedications, 20 minutes after premedications, in operating room, at anesthesia induction.
  Preoperative anxiety will be evaluated by mYPAS (modified Yale Preoperative Anxiety Scale) The mYPAS consists of 22 items in five categories (activity, emotional expressivity, state of arousal, vocalization and use of parents). The highest behavioral level observed in each of the five mYPAS categories is the score for that category. Partial weights were calculated and then added to a total score that ranged from 0 to 100. Cut off points were set to classify: a score of 23.4 to 30 for no anxiety, any score greater than 30 for anxiety.
  Change in preoperative anxiety from premedication to 20 minutes after premedication, from 20 minutes after premedication to entrance to the operating room at anesthesia induction will be evaluated.

SECONDARY OUTCOMES:
Emergence agitation | Postoperative every 10 minutes from entrance to the recovery room until discharge. If there is not a problem, patients are watched 20 minutes in our hospital's recovery room.
  Emergence agitation will be evaluated by PAED scale (pediatric anesthesia emergence delirium) The PAED scale involves five items: eye contact, purposeful actions, awareness of the surroundings, restlessness, inconsolability. First three items are scored as follows: 4= not at all, 3= just a little, 2= quite a bit, 1= very much, 0= extremely. Last two items are scored as follows: 0= not at all, 1= just a little, 2= quite a bit, 3= very much, 4= extremely. The scores of each item will summed to obtain a total score. PAED scale score of 10 or more will be defined as emergence delirium.
Mask acceptance score while mask induction | At anesthesia induction
  Anaesthesia will be induced with sevoflurane 8% and N2O 50% in oxygen by mask ventilation. The child's reaction to the mask will be evaluated by a mask acceptance scale. Mask acceptance scale to be used when assessing the child's mask acceptance is:
  1. Excellent: not scared, accepts mask easily
  2. Good: slightly scared of mask, could be calmed down easily
  3. Moderate: scared of mask, could not be calmed down
  4. Poor: crying, movement of arms and legs, struggling

CONTACTS AND LOCATIONS:
Locations (1):
- DiskapiYBERH, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Sakizci Uyar B, Polat R, Bolat M, Donmez A. Which is good for pre-operative anxiety? Midazolam, video games or teaching with cartoons: A randomised trial. Eur J Anaesthesiol. 2021 Jul 1;38(7):744-750. doi: 10.1097/EJA.0000000000001384. PMID 33186304